CLINICAL TRIAL: NCT06991569
Title: Retrospective Evaluation for Healing of Iatrogenic Perforation After Repair With Different Materials
Brief Title: Evaluation for Healing of Iatrogenic Perforation After Non Surgical Repair
Status: Completed | Type: Observational
Sponsor: Mohamed Salah Elwakeel (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Sponsor-Investigator, Mohamed Salah Elwakeel, Assistant lecturer, Ain Shams University
Organization: Ain Shams University (Other)
Other Study IDs: FDASU-REC 1117 Retrospective
Record Dates: First submitted 2025-05-09; First posted 2025-05-28 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-03

CONDITIONS: Root Perforation at the Bifurcation Area; Strip Perforation; Lateral Perforation
Keywords: Root canal perforation; Endodontics; MTA; Perforation repair material

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Non-surgical perforation repair — Root perforation repair using MTA or other perforation repair material

SUMMARY:
The goal of this retrospective study is to evaluate the outcome of nonsurgical root perforation repair treated by specialized endodontist . The null hypothesis is:

MTA can be used successfully as perforation repair material with high success rate subjects of the study were identified from patients who had received endodontic treatment with non-surgical root perforation repair by an endodontic specialist in his private practice

ELIGIBILITY:
Inclusion Criteria:

* patients who had undergone nonsurgical endodontic perforation repair

Exclusion Criteria:

* Teeth that revealed root fracture, inadequate remaining tooth structure, or severe periodontitis
* Teeth that had undergone surgical perforation repair

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: subjects were identified from among patients treated by endodontic specialist in his private clinic at Cairo, Egypt
Sampling Method: Non-Probability Sample
Enrollment: 88 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Radiographic success in terms of Healing | 7 years
  Healing outcome: the presence or absence of lesion and its size were obtained by analyzing CBCT of each case and classified into: Cases with complete resolution of lesion considered as "Healed", reduction of size considered as "Healing", and no size change or increase in lesion size considered as "Failure"

CONTACTS AND LOCATIONS:
Locations (1):
- Advanced Endodontic clinic, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided